CLINICAL TRIAL: NCT03194529
Title: Safety of FMT in Maintenance of Pediatric Crohn's Disease
Brief Title: FMT in Pediatric Crohn's Disease
Acronym: FMTPCD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHLA-17-00221
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Crohn Disease; Pediatric Crohns Disease
Keywords: Crohn's Disease; PCDAI; 16s rRNA; Fecal Microbiota Transplantation; Gut Microbiome; FMT
MeSH Terms: conditions — Crohn Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Primary outcome is safety in children with Crohn's disease in remission.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FMT in children with disease remission (Experimental): All children (with Crohn's disease in remission) will receive the equivalent of 50 g of stools from a healthy donor (FMT) into the jejunum through upper endoscopy.
  Interventions: Biological: FMT

INTERVENTIONS:
Biological: FMT — Fecal Microbiota Transplantation, single dose, 50g of stool, delivered via standard of care upper endoscopy into jejunum.
  Other Names: Fecal Microbiota Transplantation

SUMMARY:
The goal of this study is to evaluate the safety of Fecal Microbiota Transplantation (FMT) in children with Crohn's disease who are in remission. Safety will be the primary endpoint and Pediatric Crohn's Disease. Pediatric Crohn's Disease Activity Index (PCDAI) with other secondary endpoints including changes in gut microbial diversity will also be studied. All children will receive the equivalent of 50g of stools from a healthy donor into the jejunum through upper endoscopy. Also, 1-2 additional mucosal biopsies will be collected during patient's routine (standard of care) endoscopy. Subjects will have a total of 5 study visits within 24 weeks including phone call follow up on Day 7 after FMT.

DETAILED DESCRIPTION:
The Investigators hypothesize that children with Crohn's disease who are in remission can receive a single endoscopic dose of FMT with no significant safety concerns.

All children will receive the equivalent of 50 g of stools from a healthy donor into the jejunum through upper endoscopy. Children will be seen at baseline, then 4 and 24 weeks after study drug administration begins. Stools will be collected and stored for gut microbial profiles during the study visit windows. In addition, a follow up telephone call will be performed 7 days after study drug is administered. If children undergo endoscopy as part of the standard of care, study staff will obtain 1-2 additional biopsies for evaluation of mucosal inflammation. This study will also capture any laboratory results if any of the subjects undergo laboratory testing as part of the standard of care. This study will define the effects of transplant on gut microbial profile using advanced molecular taxonomic approaches. Safety will be closely monitored by solicited (during defined telephone calls and study visits) and unsolicited adverse events (at all times). Safety will be the primary endpoint of this study. Secondary endpoints include Pediatric Crohn's Disease Activity Index (PCDAI), changes in gut microbial diversity - determined by gut microbial genomics and proteomics (16S ribosomal RNA, 16s rRNA), and outcome measures for mucosal inflammation and repair as reflected through laboratory testing such as the level for C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), inflammatory cytokines of the colonic mucosa as well as the stool calprotectin level.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 7-21 who have been diagnosed with Crohn's disease
2. Remission of disease defined as PCDAI <10
3. Needs upper GI endoscopy

Exclusion Criteria:

1. Unwilling to give informed consent/assent
2. Pregnancy and breast feeding in patient subjects of childbearing potential
3. Subjects with significant renal and liver dysfunction (creatinine > 2 mg/dl and direct bilirubin > 2 mg/dl)
4. Subjects with congenital or acquired immunodeficiency, or who are immunosuppressed due to conditions other than Crohn's disease (such as neoplastic disease or organ transplantation), have received or are receiving chemotherapy, or have been diagnosed with HIV.
5. Subjects with severe food allergies

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 24 weeks
  Safety will be closely monitored (during defined telephone calls and study visits) and adverse events will be documented, including mucosal inflammation episodes and standard of care laboratory test abnormalities.

SECONDARY OUTCOMES:
Crohn's disease activity | 24 weeks
  PCDAI scores will be collected
Changes in gut microbiome | 24 weeks
  The effects of transplant on the gut microbial profile will be determined using advanced molecular taxonomic approaches (gut microbial profiling).

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Michail, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rinawi F, Assa A, Hartman C, Mozer Glassberg Y, Friedler VN, Rosenbach Y, Silbermintz A, Zevit N, Shamir R. Incidence of Bowel Surgery and Associated Risk Factors in Pediatric-Onset Crohn's Disease. Inflamm Bowel Dis. 2016 Dec;22(12):2917-2923. doi: 10.1097/MIB.0000000000000937. PMID 27755214
- [Background] Shi Y, Dong Y, Huang W, Zhu D, Mao H, Su P. Fecal Microbiota Transplantation for Ulcerative Colitis: A Systematic Review and Meta-Analysis. PLoS One. 2016 Jun 13;11(6):e0157259. doi: 10.1371/journal.pone.0157259. eCollection 2016. PMID 27295210
- [Background] Sartor RB. Microbial influences in inflammatory bowel diseases. Gastroenterology. 2008 Feb;134(2):577-94. doi: 10.1053/j.gastro.2007.11.059. PMID 18242222
- [Background] Bakhtiar SM, LeBlanc JG, Salvucci E, Ali A, Martin R, Langella P, Chatel JM, Miyoshi A, Bermudez-Humaran LG, Azevedo V. Implications of the human microbiome in inflammatory bowel diseases. FEMS Microbiol Lett. 2013 May;342(1):10-7. doi: 10.1111/1574-6968.12111. Epub 2013 Mar 15. PMID 23431991
- [Background] D'Inca R, Annese V, di Leo V, Latiano A, Quaino V, Abazia C, Vettorato MG, Sturniolo GC. Increased intestinal permeability and NOD2 variants in familial and sporadic Crohn's disease. Aliment Pharmacol Ther. 2006 May 15;23(10):1455-61. doi: 10.1111/j.1365-2036.2006.02916.x. PMID 16669960
- See also: fecal-microbial-transplant-program at CHLA — http://www.chla.org/fecal-microbial-transplant-program